CLINICAL TRIAL: NCT02913924
Title: Effect of Clonazepam on Cannabis Withdrawal and Relapse in Treatment-seeking Patients: Combined Inpatient/Outpatient Study
Brief Title: Effect of Clonazepam on Cannabis Withdrawal and Relapse in Treatment-seeking Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7343; U54DA037842-01 (NIH)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Cannabis Use Disorder
Keywords: Marijuana; Treatment
MeSH Terms: conditions — Marijuana Abuse | interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonazepam (Experimental): Clonazepam will be taken twice per day in the morning and in the evening. Clonazepam is given in a "fixed flexible" dose schedule with the dose titrated to 2mg per day or the maximum tolerated dose. Clonazepam will be taken for the first 8 weeks of the trial.
  Interventions: Drug: Clonazepam
- Placebo (Placebo Comparator): Placebo will be taken twice per day in the morning and in the evening. Placebo will be taken for the first 8 weeks of the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonazepam — fixed-flexible daily dose to a maximum of 2 mg (1 mg twice per day) for the first 8 weeks of the trial
  Other Names: Klonopin
  Arms: Clonazepam
Drug: Placebo
  Other Names: Matched Placebo
  Arms: Placebo

SUMMARY:
The proposed protocol is a double-blind, placebo-controlled inpatient and outpatient study,looking at the clinical treatment of cannabis use disorder.

The treatment study is a total of 12 weeks. There will be two options offered to participants for week 1 of the treatment study. 1) Patient will go inpatient for 5 nights and after discharge from the inpatient phase will complete the 11-weeks of outpatient treatment or 2) patients who cannot complete the inpatient phase due to work or other obligations will complete the treatment 12-week study outpatient. 80 patients seeking treatment for cannabis use disorder will be enrolled into either the inpatient/outpatient or only outpatient study. This combined design will provide a comprehensive understanding of clonazepam's effects on individuals with cannabis use disorder across a range of outcome measures while also testing the medication's ability to prevent relapse in cannabis-abstinent patients.

DETAILED DESCRIPTION:
Patients seeking treatment for Cannabis Use Disorder (CUD) will be enrolled into an inpatient laboratory for 5 nights, where they will be initiated on medication and be assessed for the influence of clonazepam (or placebo) on (1) cannabis withdrawal (mood, sleep, cannabis craving, food intake), ratings associated with medication abuse liability, cognitive performance, and (2) relapse to cannabis use after patients (now abstinent from cannabis) leave the inpatient setting maintained on clonazepam (or placebo) for 8 weeks (with a 4-week, medication-free follow up). This combined design will provide a comprehensive understanding of clonazepam's effects on individuals with cannabis use disorder across a range of outcome measures (safety, abuse liability, withdrawal symptoms) while also testing the medication's ability to prevent relapse in cannabis-abstinent patients. Patient's who are unable to complete the inpatient approach will complete the 12 week trial as an outpatient only.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM 5 criteria for CUD of at least moderate severity (≥ 4 symptoms) and is seeking treatment for cannabis use.
* Reports using cannabis a minimum of 5 days per week over the past 28 days and have positive urine test for THC on the day of study entry
* 18-65 years of age

Exclusion Criteria:

* Individuals with a lifetime DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* Individuals meeting current DSM-5 criteria for any other psychiatric disorder that may, according to the investigator's judgment, require either pharmacological or non-pharmacological intervention over the course of the study. Individuals who are currently stable on a psychotropic medication for at least 3 months may be included if in the investigator's opinion the psychotropic medication is compatible with the study medication (clonazepam). CNS depressants (e.g., benzodiazepines, opioids, adrenergic agonists) and cyp3A4 inhibitors (ketoconazole, some antipsychotics & anticonvulsants) will be exclusionary.
* Known history of allergy, intolerance or hypersensitivity to benzodiazepines
* Episodic or chronic use of benzodiazepines
* Pregnancy, lactation, or failure to use adequate contraceptive methods (condoms, diaphragm, birth control pill, IUD) in female patients who are currently engaging in sexual activity with men.
* Unstable medical conditions, such as poorly controlled hypertension, which might make participation hazardous
* Participants with a current DSM-5 diagnosis of an alcohol of substance use disorder (abuse or dependence) other than cannabis or nicotine use disorder
* Are legally mandated to participate in a substance use disorder treatment program
* Increased risk for suicide
* Current parole or probation
* Recent history of significant violent behavior
* History of current of past diagnosis of glaucoma
* History of benzodiazepine or other sedative hypnotic use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mariani, MD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- Substance Treatment Research Service (STARS) of Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo will be taken twice per day in the morning and in the evening. Placebo will be taken for the first 8 weeks of the trial.
  Placebo
Period: Overall Study
Arm/Group | Clonazepam | Placebo
Started | 34 | 34
Completed | 21 | 21
Not Completed | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonazepam | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (10.4) | 35.9 (12.0) | 35.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 3 | 17
  Not Hispanic or Latino | 20 | 31 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 16 | 29
  White | 11 | 16 | 27
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68
Marijuana Using days in prior 28 days at study start [Mean (Standard Deviation); unit: days] | 27.4 (1.5) | 27.2 (1.5) | 27.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Time to Cannabis Use Relapse
Description: for inpatient participants the number of days till relapse to cannabis use, post inpatient discharge, as recorded on the time line follow-back and confirmed by urine toxicology.
Time Frame: Number of days during 12 weeks of study participation
Population: 11 participants started the study utilizing the inpatient approach
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Clonazepam | Placebo
Number analyzed (Participants) | 6 | 5
days | 1 [0 to 1] | 1 [0 to 39]

2. Primary Outcome: Proportion of Cannabis Use Days Per Week
Description: for outpatient participants the proportion of cannabis use days per week as recorded by the Timeline Followback method
Time Frame: the 7 weeks of study participation or length of participants participation during the medication maintenance phase
Measure: Mean (Standard Deviation); unit: proportion of use days
Arm/Group | Clonazepam | Placebo
Number analyzed (Participants) | 28 | 29
proportion of use days
  week 1 | 0.74 (0.44) | 0.79 (0.41)
  week 2 | 0.78 (0.41) | 0.75 (0.44)
  week 3 | 0.71 (0.45) | 0.70 (0.46)
  week 4 | 0.67 (0.47) | 0.64 (0.48)
  week 5 | 0.67 (0.47) | 0.64 (0.48)
  week 6 | 0.58 (0.50) | 0.65 (0.48)
  week 7 | 0.58 (0.50) | 0.67 (0.47)

ADVERSE EVENTS:
Time Frame: Length of participant's participation, up to 12 weeks
Arm/Group | Clonazepam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/34
Other Adverse Events (participants affected / at risk) | 27/34 | 20/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonazepam (N=34) | Placebo (N=34)
psychotic episode (Psychiatric disorders) | 1 (1) | 0 (0)
suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonazepam (N=34) | Placebo (N=34)
insomnia (General disorders) | 2 (2) | 5 (5)
depression (Psychiatric disorders) | 2 (2) | 3 (3)
sedation (General disorders) | 10 (10) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
concentration issues (General disorders) | 2 (2) | 0 (0)
dizziness (General disorders) | 5 (5) | 2 (2)
headache (General disorders) | 4 (4) | 4 (4)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
abdominal pain (General disorders) | 0 (0) | 1 (1)
anorexia (General disorders) | 2 (2) | 1 (1)
bowel incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
dental cavities (General disorders) | 0 (0) | 1 (1)
diminished libido (General disorders) | 1 (1) | 0 (0)
erectile dysfunction (General disorders) | 1 (1) | 0 (0)
flu (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
incoordination (General disorders) | 1 (1) | 0 (0)
increased appetite (General disorders) | 0 (0) | 1 (1)
irritability (General disorders) | 2 (2) | 2 (2)
itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
memory (General disorders) | 4 (4) | 0 (0)
nightmares (General disorders) | 1 (1) | 1 (1)
orthostasis (Cardiac disorders) | 1 (1) | 0 (0)
psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
urinary incontinence (General disorders) | 2 (2) | 0 (0)
sensitivity to cannabis (General disorders) | 2 (2) | 1 (1)
palpitations (General disorders) | 1 (1) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
delayed orgasm (General disorders) | 1 (1) | 0 (0)
elevated blood pressure (Cardiac disorders) | 1 (1) | 1 (1)
drowsiness (General disorders) | 6 (6) | 2 (2)
GI upset (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
dry mouth (General disorders) | 0 (0) | 1 (1)
backache (General disorders) | 0 (0) | 1 (1)
chest discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 2 (2) | 1 (1)
mucous cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
testicular pain (General disorders) | 1 (1) | 0 (0)
confusion (General disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02913924/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT02913924/SAP_001.pdf